CLINICAL TRIAL: NCT02463071
Title: A Randomised, Double-blind, Placebo Controlled, Parallel Group, Phase III Long-term Study to Evaluate Efficacy and Safety of 12 Weeks and 52 Weeks of AZD0585 Administration, Respectively, in Japanese Patients With Hyperlipidemia Accompanied by Hypertriglyceridemia.
Brief Title: AZD0585 Phase III Long-term Study in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5884C00002
Record Dates: First submitted 2015-06-03; First posted 2015-06-04 (Estimated); Results first posted 2018-10-01 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-02

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Corn Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- AZD0585 2g group (Experimental): AZD0585 1g × 2 capsules and AZD0585 placebo 1g × 2 capsules once daily
  Interventions: Drug: AZD0585; Drug: AZD0585 placebo
- AZD0585 4g group (Experimental): AZD0585 1g × 4 capsules once daily
  Interventions: Drug: AZD0585
- Placebo control group (Placebo Comparator): AZD0585 placebo 1g × 4 capsules once daily
  Interventions: Drug: AZD0585 placebo

INTERVENTIONS:
Drug: AZD0585 — 1g soft capsule
  Other Names: Epanova
  Arms: AZD0585 2g group; AZD0585 4g group
Drug: AZD0585 placebo — 1g soft capsule
  Other Names: Corn oil
  Arms: AZD0585 2g group; Placebo control group

SUMMARY:
This study is a randomised, double-blind phase III long-term study to evaluate efficacy and safety of 12 weeks and 52 weeks of AZD0585 administration compared to placebo in patients with hyperlipidemia accompanied by hypertriglyceridemia .

ELIGIBILITY:
Key Inclusion Criteria:

* Japanese men or women, ≥20 years of age.
* Subjects must meet all of the following criteria;

  1. Fasting triglyceride level: average of Visit 2 and Visit 3 must be in the range 150 - 499 mg/dL
  2. %TG change between Visit 2 and Visit 3 must be within 30%
  3. %LDL-C change between Visit 2 and Visit 3 must be within 25%

Key Exclusion Criteria:

* Allergy or intolerance to omega-3 fatty acids and omega-3-acid ethyl esters.
* Known lipoprotein lipase impairment or deficiency, or Apolipoprotein C-II deficiency or familial dysbetalipoproteinemia.
* Current or history of pancreatitis.
* Type I diabetes mellitus, use of insulin, or haemoglobin A1c >10% at Visit 1.

Ages: 20 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2015-06-10 (Actual); Primary Completion 2017-03-11 (Actual); Study Completion 2017-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kayoko Ikeda, MD, Principal Investigator — Social medial corporation Koyokai Nakajima Hospital
Locations (22):
- Japan (22):
  - Research Site, Aki-gun
  - Research Site, Chiba
  - Research Site, Chofu-shi
  - Research Site, Fukuoka
  - Research Site, Fukuyama-shi
  - Research Site, Funabashi-shi
  - Research Site, Gifu
  - Research Site, Itami-shi
  - Research Site, Kanazawa
  - Research Site, Kawasaki-shi
  - Research Site, Koga-shi
  - Research Site, Komatsu-shi
  - Research Site, Nagoya
  - Research Site, Naha
  - Research Site, Niigata
  - Research Site, Ōta-ku
  - Research Site, Sendai
  - Research Site, Shinagawa-ku
  - Research Site, Shinjuku-ku
  - Research Site, Takamatsu
  - Research Site, Toyonaka-shi
  - Research Site, Urasoe-shi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 26 sites in Japan between 10 June 2015 and 08 March 2017.
Pre-assignment Details: The study duration was up to 60 weeks, consisting of an initial screening period of 8 weeks and a 52-week treatment period.
Period: Overall Study
Arm/Group | AZD0585 2g Group | AZD0585 4g Group | Placebo Control Group
Started | 152 | 154 | 77
Completed | 140 | 138 | 71
Not Completed | 12 | 16 | 6
Not completed — Adverse Event | 3 | 5 | 1
Not completed — Death | 1 | 0 | 0
Not completed — Eligibility criteria not fulfilled | 1 | 0 | 0
Not completed — Reason not specified | 7 | 9 | 4
Not completed — Protocol Violation | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all randomized subjects who had both baseline and any post-baseline efficacy measurements. 1 subject in Placebo group was excluded due to missing post-baseline measurements.
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD0585 2g Group | AZD0585 4g Group | Placebo Control Group | Total
Number analyzed (Participants) | 152 | 154 | 76 | 382
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.9 (10.1) | 56.5 (11.2) | 57.4 (10.9) | 56.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 29 | 13 | 83
  Male | 111 | 125 | 63 | 299
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 152 | 154 | 76 | 382
Weight [Mean (Standard Deviation); unit: kg] | 74.5 (12.8) | 75.8 (14.1) | 74.4 (13.2) | 75.0 (13.4)
BMI [Mean (Standard Deviation); unit: kg/m2] | 26.9 (4.0) | 26.9 (4.0) | 26.8 (3.9) | 26.9 (4.0)
Height [Mean (Standard Deviation); unit: cm] | 166.1 (7.8) | 167.6 (7.7) | 166.4 (9.0) | 166.8 (8.0)
Baseline triglyceride [Number; unit: Participants]
  < 300 mg/dL | 132 | 127 | 64 | 323
  >= 300 mg/dL | 20 | 27 | 12 | 59
Concurrent use of statin [Number; unit: Participants]
  Yes | 79 | 78 | 38 | 195
  No | 73 | 76 | 38 | 187
Baseline LDL-C [Number; unit: Participants]
  < 140 mg/dL | 134 | 141 | 66 | 341
  >= 140 mg/dL | 18 | 13 | 10 | 41
Baseline HDL-C [Number; unit: Participants]
  < 40 mg/dL | 43 | 52 | 22 | 117
  >= 40 mg/dL | 109 | 102 | 54 | 265
Hypertension [Number; unit: Participants]
  Yes | 97 | 103 | 44 | 244
  No | 55 | 51 | 32 | 138
Diabetes [Number; unit: Participants]
  Yes | 60 | 68 | 29 | 157
  No | 92 | 86 | 47 | 225
established CVD [Number; unit: Participants]
  Yes | 22 | 13 | 9 | 44
  No | 130 | 141 | 67 | 338

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of AZD0585 by Assessment of Percent Change in Serum Triglycerides
Description: To demonstrate the efficacy of AZD0585 2 g and 4 g compared to placebo (corn oil) in Japanese patients with hypertriglyceridemia.
Time Frame: From baseline to Week12
Population: The Full Analysis Set included all randomized patients who had both any baseline and any post-baseline efficacy measurements.
Measure: Least Squares Mean (Standard Error); unit: % (percent change from baseline)
Arm/Group | AZD0585 2g Group | AZD0585 4g Group | Placebo Control Group
Number analyzed (Participants) | 152 | 154 | 76
% (percent change from baseline) | -15.57 (1.70) | -21.78 (1.95) | 11.15 (4.65)
Statistical Analysis 1: Comparison: AZD0585 2g Group vs Placebo Control Group; Test type: Superiority; p < 0.0001, ANCOVA; Baseline TG and statin usage were included as covariates; Mean Difference (Final Values) = -26.72, 95% CI 2-sided [-36.55 to -16.88], Standard Error of Mean 4.96
Statistical Analysis 2: Comparison: AZD0585 4g Group vs Placebo Control Group; Test type: Superiority; p < 0.0001, ANCOVA; Baseline TG and statin usage were included as covariates; Mean Difference (Final Values) = -32.92, 95% CI 2-sided [-42.93 to -22.92], Standard Error of Mean 5.04

2. Primary Outcome: Safety of AZD0585 by Assessment of Adverse Events in Patients
Description: To evaluate the long-term (up to 52 weeks) safety of AZD0585 in Japanese patients with hypertriglyceridemia.
Time Frame: From baseline to Week52
Population: The Safety Analysis Set included all patients who took at least 1 dose of double-blind investigational product.
Measure: Number; unit: Participants
Arm/Group | AZD0585 2g Group | AZD0585 4g Group | Placebo Control Group
Number analyzed (Participants) | 152 | 154 | 77
Participants
  Any AE | 127 | 135 | 55
  Any AE with outcome = death | 1 | 0 | 0
  Any serious AE | 6 | 6 | 4
  Any AE leading to discontinuation of IP | 6 | 5 | 1
  Any causally related AE | 16 | 36 | 8
  Any severe AE | 4 | 1 | 0

3. Secondary Outcome: Efficacy of AZD0585 by Assessment of Percent Change in Serum Lipid Profile
Description: To assess the efficacy of AZD0585 2 g and 4 g compared to placebo (corn oil). The serum lipid profile includes total cholesterol, High-density lipoprotein cholesterol, Low-density lipoprotein cholesterol,Very low-density lipoprotein cholesterol and Non-high-density lipoprotein cholesterol.
Time Frame: From baseline to Week12
Measure: Least Squares Mean (Standard Error); unit: % (percent change from baseline)
Arm/Group | AZD0585 2g Group | AZD0585 4g Group | Placebo Control Group
Number analyzed (Participants) | 152 | 154 | 76
% (percent change from baseline)
  Total cholesterol | -0.34 (0.78) | -1.95 (1.29) | 2.31 (1.31)
  Low-density lipoprotein cholesterol | 1.45 (1.18) | -2.17 (1.91) | 2.90 (2.10)
  High-density lipoprotein cholesterol | 2.64 (0.83) | 1.54 (0.86) | 1.33 (1.22)
  Non-high-density lipoprotein cholesterol | -1.33 (1.05) | -3.11 (1.74) | 3.05 (1.83)
  Very low-density lipoprotein cholesterol | -10.18 (2.62) | -18.35 (2.73) | 7.06 (3.84)

4. Secondary Outcome: Efficacy of AZD0585 by Assessment of Percent Changes in Plasma Fatty Acids Profile.
Description: To assess the efficacy of AZD0585 2 g and 4 g compared to placebo (corn oil) . The plasma fatty acids profile includes eicosapentaenoic acid, docosahexaenoic acid, arachidonic acid and eicosapentaenoic acid per arachidonic acid rate.
Time Frame: From baseline to Week12
Measure: Least Squares Mean (Standard Error); unit: % (percent change from baseline)
Arm/Group | AZD0585 2g Group | AZD0585 4g Group | Placebo Control Group
Number analyzed (Participants) | 151 | 154 | 76
% (percent change from baseline)
  EPA | 153.06 (10.40) | 265.34 (15.86) | 3.60 (10.25)
  DHA | 14.21 (2.50) | 20.10 (2.45) | 0.13 (4.13)
  AA | -7.26 (1.33) | -10.00 (1.39) | 0.86 (1.82)
  EPA/AA ratio | 169.64 (11.12) | 319.90 (20.02) | -2.19 (9.23)

5. Secondary Outcome: Efficacy of AZD0585 by Assessment of Percent Changes in Apolipoproteins Profile
Description: To assess the efficacy of AZD0585 2 g and 4 g compared to placebo (corn oil) . Apolipoproteins include Apolipoprotein A-I, Apolipoprotein A-II, Apolipoprotein B, Apolipoprotein B48, Apolipoprotein C-II, Apolipoprotein C-III and Apolipoprotein E.
Time Frame: From baseline to Week12
Measure: Least Squares Mean (Standard Error); unit: % (percent change from baseline)
Arm/Group | AZD0585 2g Group | AZD0585 4g Group | Placebo Control Group
Number analyzed (Participants) | 151 | 154 | 76
% (percent change from baseline)
  Apo A-I | 0.39 (0.84) | -0.42 (0.83) | 0.55 (1.10)
  Apo A-II | -3.20 (0.85) | -5.01 (0.80) | 0.31 (1.01)
  Apo B | 1.73 (1.05) | -0.30 (1.07) | 2.60 (1.79)
  Apo B48 | -2.87 (4.86) | 0.94 (5.26) | 41.58 (17.49)
  Apo C-II | -2.98 (1.82) | -6.20 (2.26) | 5.49 (2.45)
  Apo C-III | -2.50 (2.03) | -5.47 (2.20) | 5.56 (2.91)
  Apo E | 5.25 (2.08) | 6.27 (2.06) | 9.67 (3.08)

6. Secondary Outcome: Efficacy of AZD0585 by Assessment of Percent Changes in Small Dense LDL and LDL-C/Apo B Ratio
Description: To assess the efficacy of AZD0585 2 g and 4 g compared to placebo (corn oil).
Time Frame: From baseline to Week12
Measure: Least Squares Mean (Standard Error); unit: % (percent change from baseline)
Arm/Group | AZD0585 2g Group | AZD0585 4g Group | Placebo Control Group
Number analyzed (Participants) | 151 | 154 | 76
% (percent change from baseline)
  Small dense LDL | -0.49 (2.08) | -1.72 (2.05) | 5.19 (2.91)
  LDL-C/Apo B ratio | 0.58 (0.99) | -1.77 (1.63) | 0.66 (1.41)

7. Secondary Outcome: Efficacy of AZD0585 by Assessment of Percent Changes in Lp(a), RLP-C, PCSK9, and Hs-CRP
Description: To assess the efficacy of AZD0585 2 g and 4 g compared to placebo (corn oil).
Time Frame: From baseline to Week12
Measure: Least Squares Mean (Standard Error); unit: % (percent change from baseline)
Arm/Group | AZD0585 2g Group | AZD0585 4g Group | Placebo Control Group
Number analyzed (Participants) | 151 | 154 | 76
% (percent change from baseline)
  Lp(a) | 14.84 (4.31) | 22.69 (3.97) | 3.18 (5.04)
  RLP-C | 5.85 (6.84) | 54.86 (55.30) | 53.80 (16.67)
  PCSK9 | 3.20 (2.79) | 0.51 (3.10) | 13.53 (4.57)
  hs-CRP | 119.94 (59.65) | 15.24 (19.29) | 69.61 (42.95)

ADVERSE EVENTS:
Time Frame: AEs, brief physical findings/clinical assessments, laboratory measurements, vital signs ,and ECGs were assessed throughout the 52-treatment period.
Arm/Group | AZD0585 2g Group | AZD0585 4g Group | Placebo Control Group
All-Cause Mortality (participants affected / at risk) | 1/152 | 0/154 | 0/77
Serious Adverse Events (participants affected / at risk) | 6/152 | 6/154 | 4/77
Other Adverse Events (participants affected / at risk) | 127/152 | 135/154 | 55/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD0585 2g Group (N=152) | AZD0585 4g Group (N=154) | Placebo Control Group (N=77)
Meningitis bacterial (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Urethral cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD0585 2g Group (N=152) | AZD0585 4g Group (N=154) | Placebo Control Group (N=77)
Bronchitis (Infections and infestations) | 11 | 12 | 5
Gastroenteritis (Infections and infestations) | 9 | 9 | 2
Influenza (Infections and infestations) | 6 | 5 | 0
Nasopharyngitis (Infections and infestations) | 56 | 56 | 28
Oral herpes (Infections and infestations) | 5 | 1 | 0
Pharyngitis (Infections and infestations) | 6 | 8 | 5
Upper respiratory tract infection (Infections and infestations) | 5 | 3 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 4 | 5 | 5
Cataract (Eye disorders) | 0 | 5 | 1
Hypertension (Vascular disorders) | 7 | 4 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Abdominal discomfort (Gastrointestinal disorders) | 4 | 6 | 0
Dental caries (Gastrointestinal disorders) | 6 | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 15 | 28 | 2
Eczema (Skin and subcutaneous tissue disorders) | 3 | 7 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 6 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 7 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-04-03): https://cdn.clinicaltrials.gov/large-docs/71/NCT02463071/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-19): https://cdn.clinicaltrials.gov/large-docs/71/NCT02463071/SAP_001.pdf